CLINICAL TRIAL: NCT04392661
Title: Female Fertility Outcome Following Bariatric Surgery: Five Years Follow up, Single Center Study
Brief Title: Female Fertility Outcome Following Bariatric Surgery: Five Years Follow up
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Shehata, Lecturer of general and pediatric surgery, Tanta University
Other Study IDs: Fertility & bariatric surgery
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Female Fertility and Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic Sleeve Gastrectomy (group I): 111 morbid obese females underwent LSG (group I). After 5 years follow up, the following were looked at: percentage excess weight loss (%EWL), comorbidity improvement or resolution, postoperative complications or mortality, fertility outcomes and breast feeding.
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy
- Laparoscopic Roux-en-Y Gastric Bypass (group II): 86 morbid obese females underwent LRYGB (group II). After 5 years follow up, the following were looked at: percentage excess weight loss (%EWL), comorbidity improvement or resolution, postoperative complications or mortality, fertility outcomes and breast feeding.
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic Sleeve Gastrectomy — bariatric surgeries and data collection
  Other Names: Laparoscopic Roux-en-Y Gastric Bypass

SUMMARY:
Maternal morbid obesity is an important risk factor in modern obstetrics, it has been associated with higher infertility rates and obstetrics complications. Bariatric surgery proven to achieve long term weight loss with improvement in all obesity related morbidities. This study was to compare the 5 years outcomes of laparoscopic sleeve gastrectomy (LSG) and laparoscopic Roux-en-Y gastric bypass (LRYGB) in terms of fertility outcomes, breast feeding, weight loss, safety, and resolution of obesity related co-morbidity.

DETAILED DESCRIPTION:
This study included 197 adult morbidly obese females, 111 underwent LSG (group I) and 86 LRYGB (group II). After 5 years follow up, the following were looked at: percentage excess weight loss (%EWL), comorbidity improvement or resolution, postoperative complications or mortality, fertility outcomes and breast feeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary goal of conceiving and complaining from infertility either primary or secondary as well as those who were seeking weight loss in preparation for marriage

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: In the LSG group, 14 patients (12.6%) suffered from infertility, and 24 patients (21.6%) were at pre-marriage stage. This is versus 15 patients (17.4%), and 26 patients (30.2%) in the LRYGB group respectively.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Measuring the number of females that got pregnant from79 females seeking pregnancy | Five years follow-up
  effect of LSG and LRYGB on female fertility and getting pregnant
percentage excess weight loss after bariatric surgery | Five years follow-up
  effect of LSG and LRYGB on percentage excess weight loss after bariatric surgery on females

SECONDARY OUTCOMES:
comorbidity improvement or resolution after bariatric surgery | Five years follow-up
  effect of LSG and LRYGB on comorbidities on females
postoperative complications or mortality after bariatric surgery | Five years follow-up
  postoperative complications or mortality after LSG and LRYGB in obese females

IPD SHARING:
Plan to Share IPD: No